CLINICAL TRIAL: NCT02615600
Title: Effectiveness of Daily Bitemporal Low-frequency Transcranial Random Noise Stimulation in Patients With Chronic Tinnitus
Brief Title: Daily Bitemporal Low-frequency Transcranial Random Noise Stimulation in Tinnitus (tRNS2-tin)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., M.D., Ph.D., University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Reg-tRNS02
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Tinnitus
Keywords: tinnitus; transcranial random noise stimulation; tRNS; auditory cortex; non-invasive brain stimulation
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lf-tRNS (Experimental): Low-frequency tRNS (Neuroconn, Eldith DC-Stimulator Plus): <100Hz, 2mA, 20min, 10s ramp time, left and right auditory cortex, 5x7cm electrode with the inferior middle part over T3/T4
  Interventions: Device: lf-tRNS

INTERVENTIONS:
Device: lf-tRNS — Low-frequency tRNS (Neuroconn, Eldith DC-Stimulator Plus): <100Hz, 2mA, 20min, 10s ramp time, left and right auditory cortex, 5x7cm electrode with the inferior middle part over T3/T4

SUMMARY:
Stimulation of the left and right auditory cortex with daily low-frequency transcranial random noise stimulation (tRNS) is used to modulate the neural pathways involved in chronic tinnitus.

DETAILED DESCRIPTION:
Tinnitus is the phantom auditory perception of sound in the absence of an external or internal acoustic stimulus. It is a frequent problem which can interfere significantly with the ability to lead a normal life. Tinnitus has been shown to be generated in the brain, as a result of functional reorganization of auditory neural pathways and the central auditory system. These changes are represented by hyper-activity and hyper-synchronicity in the auditory pathway. Treatment remains difficult. Non-invasive brain stimulation methods has shown to be effective in the treatment of chronic tinnitus with moderate effect size. First data suggest the use of transcranial random noise stimulation (tRNS) over both auditory cortices as new and highly effective treatment. Low-frequency (lf; <100Hz) tRNS might be highly effective in tackling hyper-synchronised cell assemblies. Daily lf-tRNS (2 weeks) will be examined with regard to feasibility, safety and clinical efficacy in patients suffering from chronic tinnitus in an one-arm pilot trial.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of bothersome, subjective chronic tinnitus
* diagnosis: duration of tinnitus more than 6 months

Exclusion criteria:

* objective tinnitus
* irregular head shap below the electrodes
* eczema on the head
* treatable cause of the tinnitus
* involvement in other treatments for tinnitus at the same time
* clinically relevant psychiatric comorbidity
* clinically relevant unstable internal or neurological comorbidity
* history of or evidence of significant brain malformation or neoplasm, head injury
* cerebral vascular events
* neurodegenerative disorder affecting the brain or prior brain surgery
* metal objects in and around body that can not be removed
* pregnancy
* alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
number of treatment responders | week 12
  response: tinnitus questionnaire total score reduction of at least 5 points, contrast baseline versus end of treatment (week 12)

SECONDARY OUTCOMES:
change in tinnitus questionnaire | week 2, week 4, week 12
  change in tinnitus questionnaire
change in tinnitus handicap inventory | week 2, week 4, week 12
  change in tinnitus handicap inventory
change in tinnitus numeric rating scales | week 2, week 4, week 12
  change in tinnitus numeric rating scales

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, Principal Investigator — University of Regensburg
Locations (1):
- University of Regensburg - Deptartment of Psychiatry, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No